CLINICAL TRIAL: NCT01542437
Title: Treatment With BIBW 2992, Irreversible Inhibitor of EGFR and HER-2 in Non Small Cell Lung Cancer in Advanced Stage, Which Have Progressed to Chemotherapy. Analysis of Mutations in EGFR and Number of Copies of HER-2
Brief Title: Treatment With BIBW 2992, Irreversible Inhibitor of EGFR and HER-2 in Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Principal Investigator, Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIBW2992
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Non-Small Cell Lung Cancer; EGFR; HER-2
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIBW 2992 (Experimental): Patients received a daily oral 40mg dose of afatinib. Treatment was continued until docu-mented disease progression, unacceptable toxicity or withdrawal of consent. The Common Terminology Criteria for Adverse Events (CTCAE) v4.0 was used to evaluate toxicity. In patients with severe toxicity (grade ≥3) afatinib was temporary discontinued until the patient recovery to at least grade 1 toxicity and continued with a dose reduction to 30 mg/day. Dose reduction below 30mg/day was not allowed. Patients experiencing more than one grade ≥3 event, those with grade ≥2 toxicity after dose reduction, and/or those showing no recovery within 14 days discontinued treatment.
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992 — All patients will receive: BIBW 2992 40mg every 24 hours orally, where a cycle corresponds to complete this treatment for 28 days; option 30mg/day dose reductions, according to established criteria.
  Not to be compared with any other drug.
  Other Names: Afatinib

SUMMARY:
Patients with stage IIIB and IV lung adenocarcinoma and progression to first-line chemotherapy were enrolled to receive afatinib 40 mg/day. Mutational EGFR and HER-2 status were assessed by RT-PCR. HER2 amplification was evaluated by FISH. Plasma HGF levels were measured by ELISA before and 2 months (mo) after the start of treatment. We assessed changes in serum HGF levels and their association with objective response rate (ORR), PFS and overall survival (OS).

DETAILED DESCRIPTION:
Lung cancer is the main cause of cancer-related mortality worldwide, accounting for 1.6 million deaths in 2012. Non-small-cell lung cancer (NSCLC) histology comprises ap-proximately 85% of cases. At the time of diagnosis, 75% of the patients have locally advanced or metastatic disease, with a 5-year survival rate of less than 5%. Although treatment options for these patients remain limited, drugs targeting the epidermal growth factor receptor (EGFR) have proved to be a highly effective therapy in NSCLC patients harboring sensitizing EGFR mutations.

Afatinib, a second-generation irreversible TKI, confers a theoretical advantage over re-versible TKIs in patients with acquired resistance. Through covalent binding to the kinase domain of EGFR, afatinib down regulates signaling from all homodimers and heter-odimers formed by ERBB receptor family members including EGFR, HER2 (ErbB2), HER3 (ErbB3) and HER4 (ErbB4). HER2 mutations in NSCLC are rare, being found in approximately 1-4% of lung adenocarcinomas.

In contrast with reversible TKIs, the mechanisms of resistance to irreversible TKIs have not been fully elucidated, and identification of biomarkers that predict response to these drugs, particularly in patients progressing after first line therapy, is needed. In this study we assess the usefulness of plasma HGF concentrations as a predictor of response to afatinib in patients with advanced-stage lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung cancer non-small cell (stage IIIB or IV) inoperable, locally advanced, recurrent or metastatic, histologically or cytologically documented.
* The patient must present evidence of measurable disease.
* 18 years of age or older.
* ECOG performance status of 0-2
* Life expectancy at least 12 weeks.
* lung cancer patients with advanced non-small cell, stage IIIB / IV who have received at least one cycle of systemic chemotherapy standard platinum-based first-or second-line fault has been documented that treatment.
* are admissible 3 or more prior chemotherapy regimens. Patients must have recovered from any toxic effects and should have passed at least 2 weeks after the last dose prior to registration (14 days for vinorelbine and other vinca alkaloids or gemcitabine). Patients in the opinion of the investigator are fully recovered from surgery for 4 weeks at least, can also be considered for the study. Patients must have recovered from any severe toxicity (CTC ≤ 1) caused by any previous therapy.
* granulocyte count ≥ 1.5x 109 / L and platelet count> 100 × 109 / L.
* serum bilirubin should be ≤ 1.5 X ULN
* AST and / or ALT ≤ 2 ULN (or ≤ 5 x ULN when clearly attributable to the presence of liver metastases).
* Serum creatinine ≤ 1.5 (ULN) or creatinine clearance ≥ 60ml/min
* Ability to comply with study procedures and monitoring.
* Of all women of childbearing potential should be obtained a negative pregnancy test within 72 hours before the start of therapy.
* Patients with reproductive potential must use effective contraception.
* Written informed consent (signed) to participate in the study.

Exclusion Criteria:

* Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, liver disease, renal or metabolic).
* Pre-treatment with systemic anti-tumor therapy with EGFR inhibitors (tyrosine kinase inhibitors).
* Any other malignancy within the previous 5 years (except for carcinoma in situ of the cervix or skin cancer adequately treated basal cell type).
* Excluded patients with brain metastases or spinal cord compression of newly diagnosed and / or have not been definitively treated with surgery and / or radiation, supporting both patients with CNS metastases or spinal cord compression previously diagnosed and treated with evidence of stable disease (clinically stable on imaging studies) for a minimum of 2 months.
* Any significant ophthalmologic abnormality, especially severe syndrome of dry eye, keratoconjunctivitis sicca, Sjogren's syndrome, severe keratitis exposure and any other condition that may increase the risk of corneal epithelial damage. We do not recommend the use of contact lenses during the study. The decision to continue with the use of contact lenses should be discussed with the treating oncologist and the patient's ophthalmologist.
* Patients unable to take oral medication, requiring intravenous nutrition, which have undergone prior surgical procedures affecting absorption, or who have active peptic ulceration.
* lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Overall response | from the start of consumption until at least 6 months after stopping BIBW 2992 or when all patients have died.
  Is assigned to each subject the best objective response according to the investigator's decision (according to RECIST criteria). This is defined as the best response recorded from the start of treatment until progression / recurrence of disease. For patients with response status partial (PR) or complete response (CR), changes in tumor measurements must be confirmed by repeated assessments to be made not less than 4 weeks after it first reached the response criteria The CT will be made every two months to assess response to treatment. The objective response will be summarized descriptively.
Progression Free Survival | from the start of consumption until at least 6 months after stopping BIBW 2992 or when all patients have died.
  Is defined as the time from start of treatment until the date of the first documented evidence of progression (RECIST criteria) or the date of death for any reason in the absence of disease progression (EP). For patients who have died or progressed at the time of final analysis, use the date of last contact.
Overall survival | from the start of consumption until at least 6 months after stopping BIBW 2992 or when all patients have died.
  Overall survival will be determined from the date of commencement of treatment to date of death, regardless of the cause of death. In patients who did not die at the time of final analysis will use the date of last contact.

SECONDARY OUTCOMES:
Evaluation of the HER-2 gene copy number and amplification | Baseline
  Assessing the number of copies of the HER-2 gene by FISH
DNA Extraction and Mutational Analysis of EGFR and HER-2 | Baseline
  Tumor samples were fixed in formalin and embedded in paraffin, used for histologic diagnosis of patients will be obtained from the Departments of Pathology participating institutes.
Toxicity evaluation | from the start of consumption until at least 6 months after stopping BIBW 2992 or when all patients have died.
  adverse effect from CTCAE
Determination of plasma HGF pre and post-treatment concentration | Baseline and after 2 months of treatment.
  Plasma samples were collected before the start of treatment with afatinib and after 2 months of treatment. HGF plasma levels were determined using ELISA, which was per-formed according to Quantikine human HGF immunoassay (DHG00; R&D System, Minneapolis, MN, USA). All assays were performed in duplicate. Color intensity was measured at 450 nm with a spectrophotometric plate reader. HGF concentrations were determined by comparison with standard curves.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD M Sc, Principal Investigator — Mexico. National Cancer Institute
Locations (1):
- National Cancer Institute of Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modjtahedi H, Dean C. The receptor for EGF and its ligands - expression, prognostic value and target for therapy in cancer (review). Int J Oncol. 1994 Feb;4(2):277-96. doi: 10.3892/ijo.4.2.277. PMID 21566922
- [Background] Salomon DS, Brandt R, Ciardiello F, Normanno N. Epidermal growth factor-related peptides and their receptors in human malignancies. Crit Rev Oncol Hematol. 1995 Jul;19(3):183-232. doi: 10.1016/1040-8428(94)00144-i. No abstract available. PMID 7612182
- [Background] Rusch V, Mendelsohn J, Dmitrovsky E. The epidermal growth factor receptor and its ligands as therapeutic targets in human tumors. Cytokine Growth Factor Rev. 1996 Aug;7(2):133-41. doi: 10.1016/1359-6101(96)00016-0. PMID 8899291
- [Background] Davies DE, Chamberlin SG. Targeting the epidermal growth factor receptor for therapy of carcinomas. Biochem Pharmacol. 1996 May 3;51(9):1101-10. doi: 10.1016/0006-2952(95)02232-5. PMID 8645330
- [Background] Veale D, Ashcroft T, Marsh C, Gibson GJ, Harris AL. Epidermal growth factor receptors in non-small cell lung cancer. Br J Cancer. 1987 May;55(5):513-6. doi: 10.1038/bjc.1987.104. PMID 3038157
- [Background] Sekine I, Takami S, Guang SG, Yokose T, Kodama T, Nishiwaki Y, Kinoshita M, Matsumoto H, Ogura T, Nagai K. Role of epidermal growth factor receptor overexpression, K-ras point mutation and c-myc amplification in the carcinogenesis of non-small cell lung cancer. Oncol Rep. 1998 Mar-Apr;5(2):351-4. PMID 9468555
- [Background] Pfeiffer P, Clausen PP, Andersen K, Rose C. Lack of prognostic significance of epidermal growth factor receptor and the oncoprotein p185HER-2 in patients with systemically untreated non-small-cell lung cancer: an immunohistochemical study on cryosections. Br J Cancer. 1996 Jul;74(1):86-91. doi: 10.1038/bjc.1996.320. PMID 8679464
- [Background] Cerny T, Barnes DM, Hasleton P, Barber PV, Healy K, Gullick W, Thatcher N. Expression of epidermal growth factor receptor (EGF-R) in human lung tumours. Br J Cancer. 1986 Aug;54(2):265-9. doi: 10.1038/bjc.1986.172. PMID 3017396
- [Background] Reissmann PT, Koga H, Figlin RA, Holmes EC, Slamon DJ. Amplification and overexpression of the cyclin D1 and epidermal growth factor receptor genes in non-small-cell lung cancer. Lung Cancer Study Group. J Cancer Res Clin Oncol. 1999;125(2):61-70. doi: 10.1007/s004320050243. PMID 10190311
- [Background] Fujino S, Enokibori T, Tezuka N, Asada Y, Inoue S, Kato H, Mori A. A comparison of epidermal growth factor receptor levels and other prognostic parameters in non-small cell lung cancer. Eur J Cancer. 1996 Nov;32A(12):2070-4. doi: 10.1016/s0959-8049(96)00243-2. PMID 9014747
- [Background] Fontanini G, Vignati S, Bigini D, Mussi A, Lucchi H, Angeletti CA, Pingitore R, Pepe S, Basolo F, Bevilacqua G. Epidermal growth factor receptor (EGFr) expression in non-small cell lung carcinomas correlates with metastatic involvement of hilar and mediastinal lymph nodes in the squamous subtype. Eur J Cancer. 1995;31A(2):178-83. doi: 10.1016/0959-8049(93)00421-m. PMID 7718322
- [Background] Rusch V, Baselga J, Cordon-Cardo C, Orazem J, Zaman M, Hoda S, McIntosh J, Kurie J, Dmitrovsky E. Differential expression of the epidermal growth factor receptor and its ligands in primary non-small cell lung cancers and adjacent benign lung. Cancer Res. 1993 May 15;53(10 Suppl):2379-85. PMID 7683573
- [Background] Ohsaki Y, Tanno S, Fujita Y, Toyoshima E, Fujiuchi S, Nishigaki Y, Ishida S, Nagase A, Miyokawa N, Hirata S, Kikuchi K. Epidermal growth factor receptor expression correlates with poor prognosis in non-small cell lung cancer patients with p53 overexpression. Oncol Rep. 2000 May-Jun;7(3):603-7. doi: 10.3892/or.7.3.603. PMID 10767376
- [Background] Lei W, Mayotte JE, Levitt ML. Enhancement of chemosensitivity and programmed cell death by tyrosine kinase inhibitors correlates with EGFR expression in non-small cell lung cancer cells. Anticancer Res. 1999 Jan-Feb;19(1A):221-8. PMID 10226546
- [Background] Veale D, Kerr N, Gibson GJ, Kelly PJ, Harris AL. The relationship of quantitative epidermal growth factor receptor expression in non-small cell lung cancer to long term survival. Br J Cancer. 1993 Jul;68(1):162-5. doi: 10.1038/bjc.1993.306. PMID 8391303
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Busam KJ, Capodieci P, Motzer R, Kiehn T, Phelan D, Halpern AC. Cutaneous side-effects in cancer patients treated with the antiepidermal growth factor receptor antibody C225. Br J Dermatol. 2001 Jun;144(6):1169-76. doi: 10.1046/j.1365-2133.2001.04226.x. PMID 11422037
- [Background] Van Doorn R, Kirtschig G, Scheffer E, Stoof TJ, Giaccone G. Follicular and epidermal alterations in patients treated with ZD1839 (Iressa), an inhibitor of the epidermal growth factor receptor. Br J Dermatol. 2002 Sep;147(3):598-601. doi: 10.1046/j.1365-2133.2002.04864.x. PMID 12207609
- [Background] Herbst RS, LoRusso PM, Purdom M, Ward D. Dermatologic side effects associated with gefitinib therapy: clinical experience and management. Clin Lung Cancer. 2003 May;4(6):366-9. doi: 10.3816/clc.2003.n.016. PMID 14599302
- [Background] Giovino GA. Epidemiology of tobacco use in the United States. Oncogene. 2002 Oct 21;21(48):7326-40. doi: 10.1038/sj.onc.1205808. PMID 12379876
- [Background] Li D, Ambrogio L, Shimamura T, Kubo S, Takahashi M, Chirieac LR, Padera RF, Shapiro GI, Baum A, Himmelsbach F, Rettig WJ, Meyerson M, Solca F, Greulich H, Wong KK. BIBW2992, an irreversible EGFR/HER2 inhibitor highly effective in preclinical lung cancer models. Oncogene. 2008 Aug 7;27(34):4702-11. doi: 10.1038/onc.2008.109. Epub 2008 Apr 14. PMID 18408761
- [Background] Eskens FA, Mom CH, Planting AS, Gietema JA, Amelsberg A, Huisman H, van Doorn L, Burger H, Stopfer P, Verweij J, de Vries EG. A phase I dose escalation study of BIBW 2992, an irreversible dual inhibitor of epidermal growth factor receptor 1 (EGFR) and 2 (HER2) tyrosine kinase in a 2-week on, 2-week off schedule in patients with advanced solid tumours. Br J Cancer. 2008 Jan 15;98(1):80-5. doi: 10.1038/sj.bjc.6604108. Epub 2007 Nov 20. PMID 18026190
- [Background] Yap TA, Vidal L, Adam J, Stephens P, Spicer J, Shaw H, Ang J, Temple G, Bell S, Shahidi M, Uttenreuther-Fischer M, Stopfer P, Futreal A, Calvert H, de Bono JS, Plummer R. Phase I trial of the irreversible EGFR and HER2 kinase inhibitor BIBW 2992 in patients with advanced solid tumors. J Clin Oncol. 2010 Sep 1;28(25):3965-72. doi: 10.1200/JCO.2009.26.7278. Epub 2010 Aug 2. PMID 20679611
- [Background] Sharma SV, Bell DW, Settleman J, Haber DA. Epidermal growth factor receptor mutations in lung cancer. Nat Rev Cancer. 2007 Mar;7(3):169-81. doi: 10.1038/nrc2088. PMID 17318210
- [Background] Kobayashi S, Boggon TJ, Dayaram T, Janne PA, Kocher O, Meyerson M, Johnson BE, Eck MJ, Tenen DG, Halmos B. EGFR mutation and resistance of non-small-cell lung cancer to gefitinib. N Engl J Med. 2005 Feb 24;352(8):786-92. doi: 10.1056/NEJMoa044238. PMID 15728811
- [Background] Maheswaran S, Sequist LV, Nagrath S, Ulkus L, Brannigan B, Collura CV, Inserra E, Diederichs S, Iafrate AJ, Bell DW, Digumarthy S, Muzikansky A, Irimia D, Settleman J, Tompkins RG, Lynch TJ, Toner M, Haber DA. Detection of mutations in EGFR in circulating lung-cancer cells. N Engl J Med. 2008 Jul 24;359(4):366-77. doi: 10.1056/NEJMoa0800668. Epub 2008 Jul 2. PMID 18596266
- [Background] Spicer JF, Rudman SM. EGFR inhibitors in non-small cell lung cancer (NSCLC): the emerging role of the dual irreversible EGFR/HER2 inhibitor BIBW 2992. Target Oncol. 2010 Dec;5(4):245-55. doi: 10.1007/s11523-010-0140-y. Epub 2010 Jun 24. PMID 20574858
- [Background] Takezawa K, Okamoto I, Tanizaki J, Kuwata K, Yamaguchi H, Fukuoka M, Nishio K, Nakagawa K. Enhanced anticancer effect of the combination of BIBW2992 and thymidylate synthase-targeted agents in non-small cell lung cancer with the T790M mutation of epidermal growth factor receptor. Mol Cancer Ther. 2010 Jun;9(6):1647-56. doi: 10.1158/1535-7163.MCT-09-1009. Epub 2010 Jun 8. PMID 20530710
- [Derived] Arrieta O, Cruz-Rico G, Soto-Perez-de-Celis E, Ramirez-Tirado LA, Caballe-Perez E, Martinez-Hernandez JN, Martinez-Alvarez I, Soca-Chafre G, Macedo-Perez EO, Astudillo-de la Vega H. Reduction in Hepatocyte Growth Factor Serum Levels is Associated with Improved Prognosis in Advanced Lung Adenocarcinoma Patients Treated with Afatinib: a Phase II Trial. Target Oncol. 2016 Oct;11(5):619-629. doi: 10.1007/s11523-016-0425-x. PMID 27033062